Efficacy of Wet Cupping on Reactive Oxygen Species and Antioxidant Capacity: A Self-controlled Interventional Study

## **Statistical Analysis**

Conformity to normal distribution of the data will be assessed with the Kolmogorov-Smirnov test. In groups showing normal distribution, the Student's t-test will be used in the comparison, Friedman test will be used for groups showing abnormal distribution. For paired groups showing normal distribution Paired t test, for groups showing abnormal distribution Conover test will be used. A value of p<0.05 will be accepted as statistically significant